CLINICAL TRIAL: NCT02466555
Title: The Effects of Music Therapy on Transition Outcomes in Young Adult Patients With Sickle Cell Disease
Brief Title: Music Therapy in Sickle Cell Transition Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Kulas Foundation (Other)
Responsible Party: Principal Investigator, Samuel Rodgers-Melnick, Music Therapist-Board Certified, University Hospitals Cleveland Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-15-30
Record Dates: First submitted 2015-06-04; First posted 2015-06-09 (Estimated); Results first posted 2019-09-13 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-08

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Music Therapy Group (Experimental): Music therapy is the clinical and evidence-based use of music interventions to accomplish individualized goals within a therapeutic relationship by a credentialed professional who has completed an approved music therapy program. Music therapy is an established health profession in which music is used within a therapeutic relationship to address physical, emotional, cognitive, and social needs of individuals (American Music Therapy Association [AMTA], 2013, para 1 and 2).
  Interventions: Behavioral: Music Therapy

INTERVENTIONS:
Behavioral: Music Therapy — During the educational music therapy intervention, member(s) of the Adult Sickle Cell Disease team will share with the patients the medical information pertinent to the appointment, ask health related questions of the patients and respond to any pertinent inquiries. The Music Therapist will then engage the patients and member(s) of the Adult Sickle Cell Disease team in a music therapy intervention designed to teach and reinforce the skills and knowledge presented. These music therapy interventions may include but are not limited to original songs/rap/instrumental playing, vocal and/or instrumental improvisation, patient-contributed lyrics, mnemonics, and stress and pain reducing strategies. The music therapy interventions will be tailored to best convey the educational message.

SUMMARY:
The purpose of this study is to investigate the effects of the BEATS Music Therapy Program on the self-efficacy, trust, knowledge, and adherence of young adult patients with sickle cell disease during transition.

Primary Hypotheses:

Compared to baseline, young adult patients with sickle cell disease who receive the music therapy interventions will report:

1. Higher sickle cell self-efficacy as measured by the Sickle Cell Self Efficacy Scale (SCSES),
2. Higher trust in health care providers as measured by the Wake Forest Trust in the Medical Profession Scale, and
3. Higher sickle cell disease knowledge as measured by the Seidman Sickle Cell Knowledge Quiz.

Secondary Hypotheses

1. Compared to the one year prior to the study period, young adults with sickle cell disease who receive the music therapy interventions will have a higher rate of adherence to clinic appointments during the one-year study period.

Additional Questions

1. Do music therapy interventions influence attendance to scheduled blood transfusions?
2. Do music therapy interventions influence the rate of hospital utilization as measured by Emergency Department visits, Acute Care Clinic visits, and admissions during the study period compared to the previous year?
3. Do music therapy interventions influence adherence to hydroxyurea therapy for patients receiving hydroxyurea as measured by change in mean corpuscular volume (MCV) during the study period?
4. Do music therapy interventions influence adherence to iron chelation therapy for patients receiving iron chelation therapy as measured by ferritin count during the study period?

ELIGIBILITY:
Inclusion Criteria:

* Subject is between 18 and 23 years of age
* Subject is diagnosed with sickle cell disease
* Subject is able to speak and understand English
* Subject is currently scheduled for quarterly appointments in the Bridge Clinic

Exclusion Criteria:

* Subject has significant hearing impairment that has not been corrected
* Subject has significant visual impairment that has not been corrected

Ages: 18 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-06; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel N Rodgers-Melnick, MT-BC, Principal Investigator — University Hospitals
Locations (1):
- University Hospitals Seidman Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Thirty-three participants with SCD were approached for recruitment. Three declined due to scheduling conflicts or disinterest. Thirty (90.9%) participants agreed to participate and completed written consent.
Groups:
- Music Therapy Group: Music Therapy: During the educational music therapy intervention, member(s) of the Adult Sickle Cell Disease team will share with the patients the medical information pertinent to the appointment, ask health related questions of the patients and respond to any pertinent inquiries. The Music Therapist will then engage the patients and member(s) of the Adult Sickle Cell Disease team in a music therapy intervention designed to teach and reinforce the skills and knowledge presented. These music therapy interventions may
Period: Overall Study
Arm/Group | Music Therapy Group
Started | 30
Completed | 28
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Music Therapy Group
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.04 (1.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 28
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 28
Type of Sickle Cell Disease [Count of Participants; unit: Participants]
  HbSS | 19
  HbSC | 6
  HbSBeta+ Thalassemia | 2
  HbSBeta0 Thalassemia | 1
Sickle Cell Disease Treatment [Count of Participants; unit: Participants]
  Hydroxyurea | 7
  Chronic transfusions | 9
  None | 12

OUTCOME MEASURES:

1. Primary Outcome: Change (T1 - T5) From Baseline in Scores on the Sickle Cell Self-Efficacy Scale (SCSES)
Description: Self-efficacy is the conviction that one can successfully execute the behavior required to produce the outcome. (Bandura, 1997, p. 193). The SCSES is a nine-item Likert scale originally developed for adults with sickle cell disease (Edwards, Telfair, Cecil, & Lenoci, 2000) and revised in a follow up study by Clay and Telfair (2007) for adolescents using a sample of 131 individuals age 11-19. The total score is reported with a minimum score of 9 and a maximum score of 45. Higher scores represent higher/better self-efficacy.
Time Frame: Baseline (T1), 3 months (T2), 6 months (T3), 9 months (T4), 12 months (T5), change (T1-T5) in least square mean from T1 to T5 reported
Population: All participants who participated in the music therapy intervention.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Music Therapy Group
Number analyzed (Participants) | 28
score on a scale | -1.73 [-5.55 to 2.09]

2. Primary Outcome: Change (T1-T5) From Baseline in Scores on the Wake Forest Trust in the Medical Profession Scale
Description: Patient trust is the optimistic acceptance of a vulnerable situation in which the patient believes the health-care provider will take care of the patient's interests (Dugan, Trachtenberg, & Hall, 2005).The Wake Forest Trust in the Medical Profession Scale is a five-item scale in which respondents express their level of agreement with the following statements: 1) Sometimes doctors care more about what is convenient for them than about their patients' medical needs (reverse coded); 2) Doctors are extremely thorough and careful; 3) You completely trust doctors' decisions about which medical treatments are best; 4) A doctor would never mislead you about anything; 5) All in all, you trust your doctor completely. Responses are summed and scores are on a 5-25 scale, with higher values indicating greater trust.
Time Frame: as for outcome 1
Population: All participants who participated in the music therapy intervention.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Music Therapy Group
Number analyzed (Participants) | 28
score on a scale | .18 [-2.04 to 2.39]

3. Primary Outcome: Change (T1-T5) From Baseline in Scores on the Seidman Sickle Cell Knowledge Quiz
Description: Sickle Cell Disease knowledge will be measured using the Seidman Sickle Cell Knowledge Quiz developed specifically for this study. The Seidman Sickle Cell Knowledge Quiz is adapted from questions from the Sickle Cell Disease Knowledge Test (Kaslow et al., 2000) and How Much Do I Know About Sickle Cell Disease (Baskin, Collins, Kaslow, & Hsu, 2002). The total score is reported with a minimum score of 0 and a maximum score of 12. Higher scores represent greater knowledge of sickle cell disease.
Time Frame: as for outcome 1
Population: All participants who participated in the music therapy intervention.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Music Therapy Group
Number analyzed (Participants) | 28
score on a scale | -1.88 [-2.80 to -0.97]

4. Secondary Outcome: Change From Baseline in Percentage of Attended Clinic Appointments During the One-year Study Period.
Description: Adherence is the extent to which a person's behavior coincides with medical or prescribed health advice (Julius, 2009). Adherence will be measured regularly throughout the study via medical record review. In order to assess adherence, the following data will be obtained from the medical record on each patient throughout the study period: 1) Total scheduled clinic visits with Adult Sickle Cell Disease Clinic, 2) Number of missed clinic visits to Adult Sickle Cell Disease Clinic due to no show, cancellation, or rescheduling. Adherence to clinic appointments is calculated as total number of attended clinic visits divided by total number of scheduled clinic visits (including no shows) multiplied by 100. The reported adherence percentage is the difference between percentage of visits attended during the 12 months study period minus the percentage of visits attended during the 12 months before the study period.
Time Frame: Baseline (T1), 12 months (T5)
Population: All participants who participated in the music therapy intervention.
Measure: Mean (Standard Deviation); unit: percentage of appointments attended
Arm/Group | Music Therapy Group
Number analyzed (Participants) | 28
percentage of appointments attended | 10 (40)

ADVERSE EVENTS:
Arm/Group | Music Therapy Group
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

LIMITATIONS AND CAVEATS:
Limitations to this study include missing data from some participants, lack of a control group, convenience sampling and small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes